CLINICAL TRIAL: NCT06999395
Title: Examining the Efficacy of a Multimodal Virtual Program on Pain and Sexual Outcomes in Individuals With Provoked Vestibulodynia: A Randomized Clinical Trial
Brief Title: Does a Virtual Program for Pelvic Pain Improve Pain and Sexual Outcomes in Individuals With Provoked Vestibulodynia?
Acronym: PVD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Caroline Pukall, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QueensU-196214; 196214 (Other Grant/Funding Number: Canadian Intitutes of Health Research)
Record Dates: First submitted 2025-05-09; First posted 2025-05-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Vulvodynia (Chronic Vulvar Pain); Vulvar Vestibulitis; Vestibulodynia; Provoked Vestibulodynia; Provoked Localized Vulvodynia
Keywords: vulvodynia; provoked vestibulodynia; virtual pelvic health program; pain and sexual wellbeing outcomes; randomized controlled trial; intervention
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis; Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Collaborators and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Participants in the active treatment arm will receive access to the program once determined eligible.
  Interventions: Behavioral: Virtual online pelvic health program
- Waitlist control (No Intervention): Participants in the waitlist control group will wait 3 months for access to the program. As the wait, they will receive the same surveys at the same timepoints as the active treatment group.

INTERVENTIONS:
Behavioral: Virtual online pelvic health program — The program offers a multimodal approach to self-guided treatment for PVD. Its multimodal approach is exemplified by pain education focusing on pelvic health and neuroplasticity to provide the foundation for strategies strengthening the mind-body connection to the pelvis; mindful breathing and relaxation exercises to reduce nervous system overactivation and enhance mood; and gradual progression of exercises encouraging awareness, stretching, and strengthening to promote relaxation of the pelvic floor muscles and reduction of accessory muscle tension resulting from protective guarding. The program uses 3 separate yet interconnected modules: Learn (20 modules of pain science education and skills), Rewire (11 modules featuring mindfulness and relaxation), and Move (45 pelvic and other exercises).
  Arms: Active treatment

SUMMARY:
The goal of this clinical trial is to learn if a 3-month online pelvic health program works to improve pain and sexual wellbeing in adult women with chronic genital pain. The main research questions it aims to answer are:

* How well does the program work to improve pain and sexual wellbeing?
* How well does the program work to improve pain anxiety and pain interference?
* How do participants rate their improvement after completing the program?
* How satisfied are participants with the program?

Researchers will compare participants who receive the program right away to those who wait for the program. Participants who receive the program right away will

* Progress through the program at their own pace
* Learn about pain science, do pelvic health exercises, and use information to be more mindful and less anxious about the pain
* Answer questions about their pain experiences and sexual wellbeing before and after the 3-month program, as well as 3 months after the end of the program
* Provide information about their experiences with the program and progress through the program during and after the program

DETAILED DESCRIPTION:
The primary aim of the proposed single-centre randomized controlled trial is to examine the efficacy of a virtual multimodal 12-week program for individuals with provoked vestibulodynia (PVD, diagnosed by a healthcare provider) compared with a waitlist control group (i.e., participants who are on the waitlist to receive treatment). We hypothesize that participation in the program will result in greater improvements in our primary outcomes of pain and sexual wellbeing for persons with PVD immediately post-treatment and at 3-month follow-up compared to the control group. Our secondary aim is to compare outcomes of the program versus control group on secondary measures of pain catastrophizing, pain self-efficacy, interference (on sexual life and life in general), perceived improvement, and treatment satisfaction. We hypothesize that participants in the program will report greater improvements in these outcomes compared to participants on the waitlist . We will also collect information on adverse events, progress through the program, and thoughts about the program.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported physician diagnosis of provoked vestibulodynia (PVD)
* PVD duration of at least 3 months
* PVD pain intensity rating of at least 3 on a scale from 0 (no pain) to 10 (extreme pain)
* Resides in North America (Canada or the United States)
* Fluent in English

Exclusion Criteria:

* Less than 18 years old
* Pregnancy or suspected pregnancy
* Breastfeeding
* Up to one year postpartum
* Physical or mental health conditions that significantly interfere with activities of daily living

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sexual insertional pain | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  0 (no pain) to 10 (extreme pain) rating for pain experienced during sexual activities involving vaginal insertion. Higher scores indicate higher pain intensity (worse outcomes).
Nonsexual insertional pain | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  0 (no pain) to 10 (extreme pain) rating for pain experienced during nonsexual activities involving vaginal insertion. Higher scores indicate higher pain intensity (worse outcomes).
Provoked vulvar pain by pressure/contact | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  0 (no pain) to 10 (extreme pain) rating for pain experienced during activities (sexual or nonsexual) involving pressure or contact to the vaginal opening. Higher scores indicate higher pain intensity (worse outcomes).
Sexual function | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  Female Sexual Function Index. Range of scores is 2 to 36, with higher scores indicating better sexual function (better outcomes). A score of 26.55 and lower indicates possible sexual dysfunction.
Pain interference on sexual life | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  The Sexual Function Interference subscale of the Vulvar Pain Assessment Questionnaire-Screening version will be used. Range of scores is 0-24, with higher scores indicating more interference (worse outcome).
Pain related interference on one's life | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  The activity engagement subscale of the Chronic Pain Acceptance Questionnaire (range 0-66, higher scores indicate higher levels of acceptance, which suggest better outcomes) and the Life Interference subscale of the Vulvar Pain Assessment Questionnaire-Screening version (range 0-24, higher scores indicate more interference, which suggest worse outcomes) will be used.
Participant global ratings of improvement | 12 weeks (immediate post-treatment), 3-month follow-up
  Scale of 0 (deterioration) to 5 (complete recovery) will be used. Range 0-5, with higher scores indicating more improvement.
Treatment satisfaction | 12 weeks (immediate post-treatment), 3-month follow-up
  Scale of 0 (completely dissatisfied) to 10 (completely satisfied) will be used. Range of scores, 0-10, with higher scores indicating higher treatment satisfaction.

SECONDARY OUTCOMES:
Pain Catastrophizing | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  The Pain Catastrophizing Scale will be used. Total scores range from 0-52, with higher scores indicating higher catastrophizing (worse outcomes).
Pain Self-efficacy | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  The Pain Self-Efficacy Scale will be used. Total scores range from 0-60, with higher scores indicating greater pain self-efficacy (better outcomes).
Sexual distress | Baseline, 12 weeks (immediate post-treatment), 3-month follow-up
  The 5 item Sexual Distress Scale will be used. Total scores range from 5-25, with higher scores indicating greater sexual distress (worse outcomes).

OTHER OUTCOMES:
Adverse events | At 3, 6, and 9 weeks during intervention, 12 weeks (immediate post-treatment), 3-month follow-up
  Will be collected via an open text box suitable for narrative responses from participants.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Pukall, PhD, Principal Investigator — Queen's University
Locations (1):
- Sexual Health Research Laboratory, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No